CLINICAL TRIAL: NCT05068960
Title: A Prospective Randomized Controlled Trial to Evaluate the Efficacy of an Interscalene Brachial Plexus Block and Multimodal Analgesia With and Without Liposomal Bupivacaine for Postoperative Pain Control in Total Shoulder Arthroplasty
Brief Title: Postoperative Pain Control in Total Shoulder Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scripps Clinic (Other)
Responsible Party: Principal Investigator, Heinz Hoenecke, MD, Principal Investigator, Scripps Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-19-7479
Record Dates: First submitted 2021-07-21; First posted 2021-10-06 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Total Shoulder Arthroplasty
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Double Blinded Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be blinded. Surgeon, nurses, and other clinical care providers will be blinded. Research staff will be blinded. The only staff who knows study group assignment is the pharmacist and the anesthesiologist and preoperative nurse who will administer the interscalene block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study group (Experimental): The study group will receive an interscalene block consisting of 10 mL 0.5% bupivacaine and 10 mL of liposomal bupivacaine [133mg].
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine
- Control group (Active Comparator): The control group will receive an interscalene block consisting of 20 mL of 0.5%bupivacaine alone.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Addition of liposomal bupivacaine to the interscalene block for extended pain control following total shoulder arthroplasty
  Other Names: Exparel
  Arms: Study group
Drug: Bupivacaine — Interscalene block with bupivacaine for pain control following total shoulder arthroplasty
  Other Names: Marcaine

SUMMARY:
A double blind, prospective, randomized trial to evaluate postoperative pain, narcotic use, patient satisfaction, and function among shoulder arthroplasty patients receiving interscalene block with and without the addition of liposomal bupivacaine.

DETAILED DESCRIPTION:
In order to reduce narcotic abuse potential, orthopaedic surgeons have explored multimodal pain regimens in addition to regional anesthesia to improve postoperative pain control. One commonly used intervention to reduce postoperative shoulder pain has been the interscalene brachial plexus block. This block provides significant pain relief for shoulder procedures, but has been limited to less than 24 hours even with long acting anesthetics. In the setting of shoulder arthroplasty, this short-term pain control often leads to the need for increased narcotic pain medication. Since shoulder arthroplasty has been steadily increasing in the United States with an annual growth rate of 10.6%, it is imperative to control patients' postoperative pain without increasing their risk for opiate abuse. A potential method for achieving this is by using liposomal bupivacaine in the interscalene blocks.

This study is a double blind, prospective, randomized trial to evaluate the postoperative pain profiles among shoulder arthroplasty patients receiving interscalene block with and without the addition of liposomal bupivacaine. The purpose of this study is to determine if patients undergoing shoulder arthroplasty with an interscalene brachial plexus block with liposomal bupivacaine (study group) or without liposomal bupivacaine (control group) will have differences in postoperative opiate consumption, patient-reported pain, satisfaction with surgery, and shoulder function.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing primary shoulder arthroplasty or reverse shoulder arthroplasty

Exclusion Criteria:

* Patients under the age of 50 years
* Patients over the age of 85
* Patients undergoing a revision shoulder procedure
* Documented drug or alcohol abuse
* Active narcotic use within 3 months prior to surgery
* Neurological deficit
* Allergy to amide anesthetics
* Oxycodone intolerance
* Unable to take Celebrex
* Enrollment in another clinical trial
* Comorbidity that is contraindicated with the administration of an interscalene block
* Cognitive or mental health status that interferes with study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Narcotic usage | Postoperatively (up to 1 week)
  Number and type of narcotic pain pills consumed during the first postoperative week (also converted into morphine equivalents)

SECONDARY OUTCOMES:
Severity of pain and its impact on functioning (Brief Pain Inventory - Short Form modified) | Postoperatively (at 1 week)
  Patients' self-reported pain severity and impact on functioning as measured on the Brief Pain Inventory Short-Form modified survey
Pain score (Numeric Rating Scale): Preoperatively, postoperatively, and change from preoperatively to postoperatively | Preoperatively (up to 30 days before surgery) and postoperatively (at 4 weeks), and change from preoperatively to postoperatively
  Patients' self-reported pain as measured on the Numeric Rating Scale
American Shoulder and Elbow Surgeons (ASES) score: preoperatively, postoperatively, and change from preoperatively to postoperatively | Preoperatively (up to 30 days before surgery) and postoperatively (at 4 weeks), and change from preoperatively to postoperatively
  The ASES score is a 100-point scale that evaluates two dimensions of shoulder function: pain and performance in activities of daily living. Each of the two domains make up for 50 of the 100 points. A score of 0 indicates the worst shoulder condition and a score of 100 indicates the best shoulder condition.
Satisfaction with the results of surgery (Self-Administered Patient Satisfaction Scale) | Postoperatively (at 4 weeks)
  Patients' satisfaction with results of surgery as measured on the Self-Administered Patient Satisfaction Scale
Non narcotic pain medication usage | Postoperatively (up to 1 week)
  Number and type of non-narcotic pain pills consumed during the first postoperative week

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Hoenecke, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Clinic, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No